CLINICAL TRIAL: NCT04940585
Title: Reach Out, Stay Strong, Essentials for Mothers of Newborns (ROSE), a Study of a Postpartum Depression Prevention Intervention Among Pregnant Women in a Women's Health Clinic
Brief Title: ROSE in Sunset Park
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-01961
Record Dates: First submitted 2021-04-30; First posted 2021-06-25 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Post Partum Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rose Program Group (Experimental): ROSE is a 7-session intervention. Participants will attend 6 weekly group sessions virtually, through a program on the computer called WebEx or at the clinic, and then one individual session after delivery. Participants will complete a few questionnaires at three different timepoints, including demographics, stress, social support, physical and mental health, and trauma.
  Interventions: Other: ROSE Program
- Comparison Group (No Intervention): Participants will complete three sets of questionnaires including demographics, stress, social support, physical and mental health, and trauma.

INTERVENTIONS:
Other: ROSE Program — The program includes 6 group sessions and an individual session 4-6 weeks after birth. Each session will last 60 minutes and will be conducted over Webex. The key areas that will be discussed during the sessions include: Psychoeducation, Adjusting to life with baby, Effective communication, Asking for what you need, and Planning for the future.
  Arms: Rose Program Group

SUMMARY:
The purpose of this study is to learn more about pregnant women's' experience with Reach Out, Stay Strong, Essentials for mothers of newborns (ROSE) and to evaluate the effectiveness of the ROSE program in preventing and reducing post-partum depressive symptoms, decreasing stress, and increasing social support among pregnant women.

DETAILED DESCRIPTION:
This is a 2-phase study, including a feasibility phase (Pilot, Phase 1), and an outcomes evaluation phase (Phase 2). Phase 1 tests the acceptability and feasibility of a postpartum depression prevention intervention among pregnant women attending a prenatal clinic in Sunset Park, Brooklyn. NYU research staff will be trained to implement this intervention. Based on the feedback received from women and staff in phase 1, the intervention will be modified accordingly. Phase 2 will be an outcomes evaluation to test the effectiveness of the intervention to decrease maternal stress and depressive symptoms, and increase perceived social support and self-efficacy among new mothers.

ELIGIBILITY:
Inclusion Criteria:

* Receive prenatal care at the Sunset Park Family Health Center for Women's Health and Pediatrics (SPWHP)
* Female
* At least 18 years of age
* Speaks and understands English or Spanish (depending on the language of the next group)
* Is pregnant
* Is in the second trimester of her pregnancy
* Capable of providing informed consent.
* Scores between 4 and 12 on Edinburgh Postnatal Depression Scale or records 2 or more ACEs on adapted ACEs questionnaire

Exclusion Criteria:

* Not receiving prenatal care at the Sunset Park Family Health Center for Women's Health and Pediatrics (SPWHP)
* Not female
* Under18 years of age
* Does not speak and understand English or Spanish
* Is not pregnant
* Is not in the second trimester of her pregnancy
* Is not capable of providing informed consent.
* Scoring < 4or >12 on Edinburgh Postnatal Depression Scale and scores 1 or less on adapted ACEs questionnaire.
* Positive score to #10 on the Edinburgh Postnatal Depression Scale

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 117 (Estimated)
Dates: Start 2021-03-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability of the ROSE intervention | Week 1 group session
  This will be measured by the client Satisfaction Questionnaire which is an 8-item questionnaire designed to assess the participant's satisfaction with a health service.
Acceptability of the ROSE intervention | Week 2 group session
  This will be measured by the client Satisfaction Questionnaire which is an 8-item questionnaire designed to assess the participant's satisfaction with a health service.
Acceptability of the ROSE intervention | Week 3 group session
  This will be measured by the client Satisfaction Questionnaire which is an 8-item questionnaire designed to assess the participant's satisfaction with a health service.
Acceptability of the ROSE intervention | Week 4 group session
  This will be measured by the client Satisfaction Questionnaire which is an 8-item questionnaire designed to assess the participant's satisfaction with a health service.
Acceptability of the ROSE intervention | Week 5 group session
  This will be measured by the client Satisfaction Questionnaire which is an 8-item questionnaire designed to assess the participant's satisfaction with a health service.
Acceptability of the ROSE intervention | Week 6 group session
  This will be measured by the client Satisfaction Questionnaire which is an 8-item questionnaire designed to assess the participant's satisfaction with a health service.
Acceptability of the ROSE intervention | Post-birth Visit (4-5 weeks after birth)
  This will be measured by the client Satisfaction Questionnaire which is an 8-item questionnaire designed to assess the participant's satisfaction with a health service.
Change in level of postpartum depression | Baseline Visit, Week 1 group session, Week 2 group session, Week 3 group session, Week 4 group session, Week 5 group session,Week 6 group session,, Post-birth Visit (4-5 weeks after birth)
  This will be measured by the Edinburgh Postnatal Depression Scale (EPDS) which is a 10-item questionnaire. Mothers are asked to answer each question in terms of the past seven days. Mothers scoring above 12 or 13 are likely to be suffering from depression and should seek medical attention.

SECONDARY OUTCOMES:
Change in the level of self-efficacy | Baseline Visit, Week 1 group session, Week 2 group session, Week 3 group session, Week 4 group session, Week 5 group session,Week 6 group session,, Post-birth Visit (4-5 weeks after birth)
  This will be measured by using the General Self-Efficacy Scale (GSE). The General Self-Efficacy Scale is a 10-item psychometric scale that is designed to assess optimistic self-beliefs to cope with a variety of difficult demands in life.
Change in perceived social support | Baseline Visit, Week 1 group session, Week 2 group session, Week 3 group session, Week 4 group session, Week 5 group session,Week 6 group session,, Post-birth Visit (4-5 weeks after birth)
  The Multidimensional Scale of Perceived Social Support (MSPSS) is a brief questionnaire designed to measure perceptions of support from 3 sources: Family, Friends, and a Significant Other. The scale is comprised of a total of 12 items, with 4 items for each subscale.
Change in perception of stress | Baseline Visit, Week 1 group session, Week 2 group session, Week 3 group session, Week 4 group session, Week 5 group session,Week 6 group session,, Post-birth Visit (4-5 weeks after birth)
  The Perceived Stress Scale (PSS) is the most widely used psychological instrument for measuring the perception of stress. It is a measure of the degree to which situations in one's life are appraised as stressful. The scale also includes a number of direct queries about current levels of experienced stress.

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Kerker, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request